CLINICAL TRIAL: NCT05468086
Title: Effects of Virtual Reality on Pain and Anxiety Using Validated Surveys and Biodata Analysis
Brief Title: VR Solace for Pain and Anxiety Using Survey and Biodata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Liran (Other)
Responsible Party: Sponsor-Investigator, Omer Liran, Assistant Professor, Department of Psychiatry & Behavioral Neurosciences, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002144
Record Dates: First submitted 2022-07-13; First posted 2022-07-21 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Solace VR (Experimental): This arm will include software that provides immersive distraction based content for pain reduction.
  Interventions: Device: VR Solace

INTERVENTIONS:
Device: VR Solace — Participants will use the VR audio and visual head-mounted device. The device is a standalone VR headset. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view.

SUMMARY:
The purpose of this study is to assess the therapeutic response to VR Solace in patients with chronic pain and anxiety using real-time clinical and survey data. Regression analysis of demographic characteristics, lab and survey data will be conducted to better understand the efficacy of VR Solace in treating chronic pain and anxiety. The investigator also aims to explore the possible association between the patient-reported changes in pain or anxiety levels with real-time physiological changes observed during VR Solace use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Endorsing pain/anxiety with objective measurement of 3 or greater on 10-point scale on validated survey
* Diagnosis with chronic pain/anxiety

Exclusion Criteria:

* Exclusion of patients that are followed by CL Psychiatry team at Cedars-Sinai Medical Center to avoid overlap with another ongoing VR study
* No active diagnosis of medical conditions that may cause physiological variations in vital signs (i.e. sepsis, cardiogenic shock/arrhythmia)
* No active diagnosis of seizures, migraines, severe nausea, severe propensity for motion sickness, or facial/head deformities that would allow for comfortable placement of headset
* Exclusions of patient currently taking beta blockers
* Unable to communicate/read English for survey items
* Unable to use VR independently - patients will be expected to maneuver through questions/steps of the VR system during the session

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Liran, MD, MSHS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment will be limited to one site, an inpatient hospital setting at Cedars-Sinai Medical Center (CSMC)
Period: Overall Study
Arm/Group | Solace VR
Started | 35
Completed | 31
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Subject was found ineligible after consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Solace VR
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Pain Level Pre Versus Post-VR Session
Description: Pain level pre- versus post-VR Solace as measured by Patient-Reported 11-point numeric rating scale (Continuous, 0-10, higher the worse).
Time Frame: Just prior to session to 15-minutes post session
Population: Age 18 years or older who suffer from chronic pain, have ongoing pain of equal or greater than 3 on an 11-point numerical rating scale, and were capable of giving informed consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-Solace VR: This arm is participants pre-VR intervention
  VR Solace: Participants will use the VR audio and visual head-mounted device. The device is a standalone VR headset. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view.
- Post-VR Solace: This arm is participants post-VR intervention
Arm/Group | Pre-Solace VR | Post-VR Solace
Number analyzed (Participants) | 31 | 31
score on a scale | 6.6 (2.0) | 5.1 (2.5)

2. Primary Outcome: Patient-reported Anxiety Level Pre Versus Post-VR Session
Description: Anxiety level pre versus post-VR Solace as measured by Patient-Reported 6-question version of State-Trait Anxiety Inventory (4-point scale, 1 to 4, for each question, e.g. from "Almost Never" to "Almost Always". The scores are added up to produce a total score of anxiety. Higher scores indicate greater anxiety). Scores range from 20 to 80, with higher scores reflecting increased anxiety.
Time Frame: Just prior to VR session and 15 minutes after the VR session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-Solace VR: This is pre- software that provides immersive distraction based content for pain reduction.
  VR Solace: Participants will use the VR audio and visual head-mounted device. The device is a standalone VR headset. The device supports 3 degrees of freedom (3DOF) head tracking, has best-in-class optics, and a wide field-of-view.
- Post-VR Solace: This is post- software that provides immersive distraction based content for pain reduction.
Arm/Group | Pre-Solace VR | Post-VR Solace
Number analyzed (Participants) | 31 | 31
score on a scale | 46.7 (12.2) | 35.6 (11.2)

ADVERSE EVENTS:
Time Frame: Up to 15 minutes post-VR session
Description: Adverse events were collected by interview post VR session. There were no adverse events reported.
Arm/Group | Solace VR
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT05468086/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT05468086/ICF_001.pdf